CLINICAL TRIAL: NCT03196089
Title: Effect of Short-term Oxygen Therapy on Cardiopulmonary Exercise (CPET) Capacity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Short-term Oxygen During CPET in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KEK-ZH-NR. 2012-0251_2
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental oxygen (Experimental): Supplemental oxygen will be applied via a mask during CPET
  Interventions: Procedure: Oxygen application
- Sham room air (Sham Comparator): Room air will be applied similarly to oxygen
  Interventions: Procedure: Oxygen application

INTERVENTIONS:
Procedure: Oxygen application — Supplemental oxygen via mask

SUMMARY:
In a randomized, sham-controlled trial the investigators will test whether supplemental oxygen given during cardiopulmonary exercise testing will improve exercise performance and physiological parameters in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic obstructive pulmonary disease
* on optimized medical therapy and in stable condition for at least 4 week
* desaturate in the 6 minute walking test by at least 4% to values <92%

Exclusion Criteria:

* unstable conditions
* pregnant women
* patients with relevant concomitant lung disease and severe daytime hypoxemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Watt | 1 day
Exercise time | 1 day

SECONDARY OUTCOMES:
Peak Oxygen uptake | 1 day
Respiratory Exchange ratio | 1 day
Ventilatory equivalent of carbon dioxide (VE/VCO2) slope | 1 day
End-tidal pressures of carbon dioxide (PET CO2) | 1 day
Changes in arterial blood parameters | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, Prof. Dr., Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No